CLINICAL TRIAL: NCT04142021
Title: A Multicenter, Pilot Study to Evaluate Safety and Feasibility Evaluation of Planning and Execution of Surgical Revascularization Solely Based on Coronary CTA and FFRCT in Patients With Complex Coronary Artery Disease (FASTTRACK CABG)
Brief Title: Safety and Feasibility Evaluation of Planning and Execution of Surgical Revascularization Solely Based on Coronary CTA and FFRCT in Patients With Complex Coronary Artery Disease (FASTTRACK CABG)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: GE Healthcare (Industry); HeartFlow, Inc. (Industry)
Responsible Party: Principal Investigator, Patrick Serruys, Professor / Chairman of the study, National University of Ireland, Galway, Ireland
Other Study IDs: FASTTRACK CABG
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: coronary artery bypass graft; coronary computed tomography angiography; fractional flow reserve derived from computed tomography angiography; invasive coronary angiography, revascularization
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with 3-vessel disease with or without left main: Patients with 3-vessel disease with or without left main involvement referred to CABG treatment based on coronary angiography.
  Interventions: Diagnostic Test: Coronary computed tomography angiography

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography — Surgery planning done based solely on coronary computed tomography angiography.

SUMMARY:
To assess the feasibility of coronary computed tomography angiography (CTA) and fractional flow reserve derived from CTA (FFRCT) to replace invasive coronary angiography (ICA) as a surgical guidance method for planning and execution of coronary artery bypass graft (CABG) in patients with 3-vessel disease with or without left main disease. The FASTTRACK CABG study is an investigator-initiated single-arm, multicentre, prospective, proof-of-concept, and first-in-man study with feasibility and safety analysis. Surgical revascularization strategy and treatment planning will be solely based on coronary CTA and FFRCT without knowledge of the anatomy defined otherwise by ICA that will be viewed and analyzed only by the conventional heart team. Clinical follow-up visit including coronary CTA will be performed 30 days after CABG in order to assess graft patency and adequacy of the revascularization with respect to the surgical planning based on non-invasive imaging with functional assessment and compared to ICA. Primary feasibility endpoint is CABG planning and execution solely based on coronary CTA in 114 patients. Primary safety endpoint based on 30-day coronary CTA is graft assessment either at the ostium, in the shaft or at the anastomoses of each individual graft either single or sequential. The FASTTRACK CABG study is the first study to assess safety and feasibility of planning and execution of surgical revascularization in patients with complex coronary artery disease, solely based on coronary CTA combined with FFRCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to CABG treatment (as assessed by 'conventional heart team') having at the time of the conventional heart team evaluation at least 1 de novo stenotic lesion (with a visually assessed DS with ≥ 50%) in all 3 major epicardial territories [left anterior descending (LAD) and/or side branch, left circumflex artery (LCX) and/or side branch, right coronary artery (RCA) and/or side branch] supplying viable myocardium with or without left main involvement
* Patients with hypoplastic RCA with absence of descending posterior and presence of a lesion in the LAD and LCX territories may be included in the trial as a 3VD equivalent. Ostial LAD plus ostial LCX may be included in the trial as a left main equivalent
* Distal vessel size should be at least 1.5 mm in diameter as visually assessed in the diagnostic angiogram (as requested by the surgeons)
* Patients with silent ischemia, chronic coronary syndrome or stabilized acute coronary syndrome with normalized (stable or decreasing) cardiac biomarker values. For patients showing elevated troponin (cTn) (e.g. non-ST elevation myocardial infarction [NSTEMI] patients) at baseline (within 24h pre-CABG) an additional blood sample must be collected prior to CABG to confirm that: a) hs-cTn or troponin I or T levels are stable, i.e. the value should be within 20% range of the value found in the first sample at baseline, or have dropped 25; b) creatine kinase-muscle/brain (CK-MB) and creatine kinase (CK) levels are within normal range. If hs-cTn or troponin I or T levels are stable or have dropped, or the CK-MB and CK levels are within normal ranges and the ECG is normal, patients may be included in the study
* All anatomical SYNTAX Scores are eligible
* Patients are amenable to coronary CTA (e.g. no claustrophobia, high heart rate not amenable to beta-blockers, poor renal function, etc., up to the discretion of the investigator)
* Patients have been informed of the nature of the study and agree to its provisions and have provided written informed consent as approved by the Ethical Committee of the respective clinical site
* Patients agree to 1-month follow-up visit including coronary CTA

Exclusion Criteria:

* Under the age of 18 years
* Unable to give informed consent
* Known pregnancy at the time of enrollment; female of childbearing potential, i.e. who are not surgically sterile or post-menopausal (defined as no menses for 2 years without an alternative cause); female who is breastfeeding at time of enrollment
* Prior PCI or CABG; history of coronary stent implantation
* Evidence of evolving or ongoing ST-elevation MI (STEMI) on ECG and/or elevated cardiac biomarkers (according to local standard hospital practice) have not returned within normal limits at the time of enrollment (non-STEMI)
* Known renal insufficiency (e.g. serum creatinine >2.5mg/dL, or creatinine clearance ≤30 mL/min), or need for dialysis, or acute kidney failure (as per physician judgment)
* Concomitant cardiac valve disease requiring surgical therapy (repair or replacement) and/or aneurysmectomy
* Single or two-vessel disease (at time of the conventional heart team consensus)
* Non-graftable distal bed in >1 vessel as assessed by the surgeon based on ICA
* Persistent atrial fibrillation or significant arrhythmias
* Known allergy to iodinated contrast
* A body mass index (BMI) of 35 or greater
* Currently participating in another clinical trial not yet at its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 3-vessel disease with or without left main involvement referred to CABG treatment.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility expressed in percentage of CABG planning and execution solely based on coronary CTA in 114 candidates for CABG (i.e. the 'CTA heart team' and the operator being blind for the ICA). [percentage/rate]. | 2 weeks after enrollment
Safety: The rate of graft stenosis [≥ 50% diameter stenosis (DS) - 99% DS] or occlusion (100% DS) either at the ostium, in the shaft or at the level of the sequential anastomosis or at the distal anastomosis of each individual graft based on coronary CTA | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital of Brussels, Brussels, Belgium
- University Hospital of Jena, Jena, Germany
- Centro Cardiologico Monzino, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The research data will be entered on separate forms and stored under a code number, according to prevailing legal requirements. No names or other personal data will be stored. Only the study doctor will hold the information to link the code to the patients. The encoded data will be processed, analysed and reported by the research employees of this study, who have an obligation of secrecy.
  Representatives of the sponsor or members of the Ethics Committee (EC) and regulatory authorities within Europe can have access to the medical files in order to inspect the correctness of the research data. Data may be provided to representatives and affiliates of the industries supporting the study: General Electric and HeartFlow Inc. It is possible that the results of this study are presented or published in medical journals; this will always be without mention of the identity of the patients.

REFERENCES:
- [Derived] Revaiah PC, Tsai TY, Farina J, Ferraz-Costa G, Jongenotter J, Oshima A, Garg S, Puskas JD, Narula J, Gupta H, Agarwal V, Tanaka K, De Mey J, La Meir M, Schneider U, Kirov H, Saima M, Teichgraber U, Pompilio G, Pontone G, Andreini D, Morel MA, Doenst T, Onuma Y, Serruys PW. High-risk plaques in proximal and distal segments relative to graft anastomoses and non-grafted segments. J Cardiovasc Comput Tomogr. 2025 Nov-Dec;19(6):684-693. doi: 10.1016/j.jcct.2025.09.013. Epub 2025 Oct 9. PMID 41068029
- [Derived] Miyashita K, Onuma Y, Oshima A, Tobe A, Tsai TY, Revaiah PC, Tu S, Reiber JHC, Andreini D, Mushtaq S, Pontone G, Pompilio G, De Mey J, Tanaka K, La Meir M, Kirov H, Doenst T, Teichgraber U, Narula J, Puskas JD, Gupta H, Garg S, Serruys PW. Fractional flow reserve from coronary CT angiography compared with quantitative flow ratio in complex CAD. J Cardiovasc Comput Tomogr. 2025 Nov-Dec;19(6):701-710. doi: 10.1016/j.jcct.2025.09.001. Epub 2025 Sep 22. PMID 40983565
- [Derived] Masuda S, Revaiah PC, Kageyama S, Tsai TY, Miyashita K, Tobe A, Puskas JD, Teichgraber U, Schneider U, Doenst T, Tanaka K, De Mey J, La Meir M, Mushtaq S, Bartorelli AL, Pompilio G, Garg S, Andreini D, Onuma Y, Serruys PW. Quantitative coronary computed tomography assessment for differentiating between total occlusions and severe stenoses. J Cardiovasc Comput Tomogr. 2024 Sep-Oct;18(5):450-456. doi: 10.1016/j.jcct.2024.04.013. Epub 2024 May 7. PMID 38714459
- [Derived] Serruys PW, Kageyama S, Pompilio G, Andreini D, Pontone G, Mushtaq S, La Meir M, De Mey J, Tanaka K, Doenst T, Teichgraber U, Schneider U, Puskas JD, Narula J, Gupta H, Agarwal V, Leipsic J, Masuda S, Kotoku N, Tsai TY, Garg S, Morel MA, Onuma Y. Coronary bypass surgery guided by computed tomography in a low-risk population. Eur Heart J. 2024 May 27;45(20):1804-1815. doi: 10.1093/eurheartj/ehae199. PMID 38583086
- [Derived] Kawashima H, Pompilio G, Andreini D, Bartorelli AL, Mushtaq S, Ferrari E, Maisano F, Buechel RR, Tanaka K, La Meir M, De Mey J, Schneider U, Doenst T, Teichgraber U, Stone GW, Sharif F, de Winter R, Thomsen B, Taylor C, Rogers C, Leipsic J, Wijns W, Onuma Y, Serruys PW. Safety and feasibility evaluation of planning and execution of surgical revascularisation solely based on coronary CTA and FFRCT in patients with complex coronary artery disease: study protocol of the FASTTRACK CABG study. BMJ Open. 2020 Dec 10;10(12):e038152. doi: 10.1136/bmjopen-2020-038152. PMID 33303435